CLINICAL TRIAL: NCT03006237
Title: A Phase 1 Open Label Single Center Safety, Tolerability and Pharmacokinetic Study of IS-001 Injection in Patients Undergoing Robotic Hysterectomy Using the da Vinci® Si/Xi Surgical System With Firefly® Fluorescent Imaging
Brief Title: IS-001 Injection Phase-1 Safety, Tolerance and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISI-001-01
Record Dates: First submitted 2016-12-14; First posted 2016-12-30 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Hysterectomy; Surgery
MeSH Terms: interventions — IS 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV IS-001 drug (Experimental): IV IS-001 given during hysterectomy performed with da Vinci® Si/Xi Surgical System
  Interventions: Drug: IS-001; Device: da Vinci® Si/Xi Surgical System

INTERVENTIONS:
Drug: IS-001 — 10mg, 20mg or 40 mg IV IS-001 drug administered during surgery
Device: da Vinci® Si/Xi Surgical System — robot-assisted minimally invasive hysterectomy surgery performed with da Vinci® Si/Xi Surgical System with Firefly® Fluorescent Imaging

SUMMARY:
A Phase 1 Open Label Single Center Safety, Tolerability and Pharmacokinetic Study of IS-001

DETAILED DESCRIPTION:
A Phase 1 Open Label Single Center Safety, Tolerability and Pharmacokinetic Study of IS-001 Injection in Patients Undergoing Robotic Hysterectomy Using the da Vinci® Si/Xi Surgical System with Firefly® Fluorescent Imaging

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 18 and 65.
2. Subject is scheduled to undergo robotic hysterectomy using a da Vinci® Si/Xi surgical system with Firefly® fluorescent imaging.
3. Subject is willing and able to provide informed consent.
4. Subject is considered capable of complying with study procedures.
5. Subject has no medical history of liver or kidney disease.
6. Subject has no evidence of NYHA Class II-IV cardiac disease.
7. Subject has recent (< 3 months) clinical hematology (CBC) values within the acceptable values reference range.
8. Subject has recent (< 3 months) clinical serum chemistry (CMP) values within the acceptable values reference range.

Exclusion Criteria:

1. Subject is pregnant or nursing.
2. Subject has a history of alcoholism.
3. Subject has a history of drug abuse.
4. Subject has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
5. Subject has known human immunodeficiency virus (HIV) infection.
6. Subject has been diagnosed with or treated for cancer in the last 2 years.
7. Subject has a total body weight < 32 kg.
8. Subject has after 5 minutes of supine rest a diastolic blood pressure ≥100 mmHg and/or a systolic blood pressure ≥160 mmHg.
9. Subject has after 5 minutes of supine rest a resting heart rate ≤35 or ≥115 bpm.
10. Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data or represents an unacceptable safety liability.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Monitor Safety Parameters (vital signs, ECG, serum chemistry and hematology, urinalysis and adverse events) | 14 days
  Vital signs, 12-lead ECG, serum chemistry (CMP) and hematology (CBC), urinalysis and incidence of treatment-emergent adverse events

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of IS-001: Cmax | 6 hours
  Pharmacokinetics for IS-001 as measured by maximum serum/drug concentration
Evaluation of pharmacokinetic parameter of IS-001: Tmax | 6 hours
  Pharmacokinetics for IS-001 as measured by the time to maximum serum/drug concentration
Evaluation of pharmacokinetic parameter of IS-001: t1/2 | 6 hours
  Pharmacokinetics for IS-001 as measured by terminal elimination half-life
Evaluation of pharmacokinetic parameter of IS-001: AUC | 6 hours
  Pharmacokinetics for IS-001 as measured by area under the serum/drug concentration time curve

CONTACTS AND LOCATIONS:
Overall Officials: Richard Farnam, MD, Principal Investigator — Texas Urogynecology and Laser Surgery Center, Las Palmas Medical Center
Locations (1):
- Las Palmas Medical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farnam RW, Arms RG, Klaassen AH, Sorger JM. Intraoperative ureter visualization using a near-infrared imaging agent. J Biomed Opt. 2019 Jun;24(6):1-8. doi: 10.1117/1.JBO.24.6.066004. PMID 31215195